CLINICAL TRIAL: NCT01223755
Title: EFFECTS OF SIROLIMUS ON DISEASE PROGRESSION IN PATIENTS WITH AUTOSOMAL DOMINANT POLYCYSTIC KIDNEY DISEASE AND SEVERE RENAL INSUFFICIENCY
Brief Title: Sirolimus In Autosomal Dominant Polycystic Kidney Disease And Severe Renal Insufficiency
Acronym: SIRENA-II
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: safety and efficacy reason
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRENA-II; 2007-005047-21 (EudraCT Number)
Record Dates: First submitted 2010-10-12; First posted 2010-10-19 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Autosomal dominant polycystic kidney disease; Sirolimus; Renal insufficiency
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Renal Insufficiency | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Experimental)
  Interventions: Drug: Sirolimus
- conventional therapy (Active Comparator)
  Interventions: Drug: conventional therapy

INTERVENTIONS:
Drug: Sirolimus — Patients will be given SRL for one year starting at the oral daily dose of 3 mg, with periodical whole blood level measurements. The daily dose will be adjusted to keep SRL concentration within 5-10 ng/ml. Drug levels will be assessed at day 7 after starting treatment and every two weeks for the first month. Subsequently SRL concentrations will be monitored at monthly intervals (or at least 5 days after drug dose adjustments) until the end of the treatment period.
  Other Names: Rapamune
  Arms: Sirolimus
Drug: conventional therapy — Conventional treatment relates usually to the administration of antihypertensive drugs for patients with high blood pressure. Thus, for the present study, no major change in antihypertensive treatment should be introduced throughout the whole study period unless deemed clinically necessary (the reasons of the changes should be, however, clearly explained in the CRF). Only small changes in the doses of the ongoing treatments are recommended in order to maintain the same level of blood pressure control (target systolic/diastolic blood pressure <130/80 mmHg). This approach is aimed to minimize the confounding effect of any change in concomitant treatments on some efficacy variables (such as urinary protein excretion rate).
  Arms: conventional therapy

SUMMARY:
The general aim of this study in adult patients with Autosomal Dominant Polycystic Kidney Disease (ADPKD) and severe renal insufficiency is to assess the safety and the efficacy of sirolimus (SRL) in slowing renal function decline as compared to conventional therapy.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common hereditary renal disease, responsible for the 8% to 10% of the cases of end-stage renal disease (ESRD) in Western Countries.

ADPKD shows genetic heterogeneity, with at least three different genes implicated: the PKD1 gene (85% of the cases), the PKD2 (15% of the cases), and probably a PDK3 gene not yet identified. Recently, it has been reported that PC1 tail interacts with tuberin, the product of the TSC2 gene. The main function of the tuberin is to inactivate the Ser/Thr kinase mTOR, whose activity has been linked to increased cell growth, proliferation, apoptosis and differentiation. In ADPKD experimental animal models, researchers have shown that cyst lining epithelial cells exhibited very high mTOR activity; thus, they hypothesized that PC1 normally suppresses mTOR activity, and that defects in PC1 (and other proteins) may lead to aberrant mTOR activation. Studies in rat models of ADPKD have shown that short-term treatment with sirolimus (SRL) resulted in the dramatic reduction of the kidney size.

Recently we have documented that in ADPKD patients with normal kidney function or moderate renal dysfunction a short-course of SRL halted cyst growth and increased parenchyma volume. At this effective SRL dose (target trough blood level 5-10 ng/ml) the only relevant adverse effect observed in some patients was the development of aphthous stomatitis, relieved with topical treatment alone using a mouthwash.

Interestingly a retrospective study in a small number of SRL-treated ADPKD transplant patients showed that the treatment significantly reduced native kidney volumes over an average of 24 month follow-up. This reduction was three times higher than that reported in a control group of ADPKD transplant recipients not given SRL over a 40 month period. These results suggested that SRL may have a similar beneficial effect in humans as in experimental animals.

Overall, these findings are the basis for designing this study in ADPKD patients with severe renal dysfunction (GFR 40-15 ml/min/1.73m2) aimed to assess the safety and the efficacy of SRL in slowing renal function decline as compared to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical and ultrasound diagnosis of ADPKD
* GFR 40-15 ml/min/1.73 m2 (estimated by the 4 variable MDRD equation)
* Urinary protein excretion rate < 0.5 g/ 24 hrs
* Written informed consent

Exclusion Criteria:

* Diabetes
* Urinary protein excretion rate >0.5 g/ 24 hrs or abnormal urinalysis suggestive of concomitant, clinically significant glomerular disease
* Urinary tract lithiasis, infection or obstruction
* Cancer
* Psychiatric disorders and any condition that might prevent full comprehension of the purposes and risks of the study
* Pregnancy, lactation or child bearing potential and ineffective contraception (estrogen therapy in post menopausal women should not be stopped)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) | At baseline.
  To compare changes over baseline of GFR (delta GFR) measured by plasma iohexol clearance in SRL and conventional treatment ADPKD patients.
Glomerular Filtration Rate (GFR) | At 12th month .
  To compare changes over baseline of GFR (delta GFR) measured by plasma iohexol clearance in SRL and conventional treatment ADPKD patients.
Glomerular Filtration Rate (GFR) | After six months from baseline.
  To compare changes over baseline of GFR (delta GFR) measured by plasma iohexol clearance in SRL and conventional treatment ADPKD patients.
Glomerular Filtration Rate (GFR) | Every 12 months.
  To compare changes over baseline of GFR (delta GFR) measured by plasma iohexol clearance in SRL and conventional treatment ADPKD patients.

SECONDARY OUTCOMES:
Liver volume parameters. | At baseline.
  To compare absolute and relative changes over baseline of liver volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.
Renal volume parameters. | At baseline.
  To compare absolute and relative changes over baseline of renal volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.
Liver volume parameters. | At 12 month.
  To compare absolute and relative changes over baseline of liver volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.
Liver volume parameters. | At 36 month.
  To compare absolute and relative changes over baseline of liver volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.
Renal volume parameters. | At 12 month.
  To compare absolute and relative changes over baseline of renal volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.
Renal volume parameters. | At 36 month.
  To compare absolute and relative changes over baseline of renal volume parameters, assessed by contrast-enhanced spiral computed tomography, in SRL and conventional treatment ADPKD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Negri Institute - Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Ruggenenti P, Gentile G, Perico N, Perna A, Barcella L, Trillini M, Cortinovis M, Ferrer Siles CP, Reyes Loaeza JA, Aparicio MC, Fasolini G, Gaspari F, Martinetti D, Carrara F, Rubis N, Prandini S, Caroli A, Sharma K, Antiga L, Remuzzi A, Remuzzi G; SIRENA 2 Study Group. Effect of Sirolimus on Disease Progression in Patients with Autosomal Dominant Polycystic Kidney Disease and CKD Stages 3b-4. Clin J Am Soc Nephrol. 2016 May 6;11(5):785-794. doi: 10.2215/CJN.09900915. Epub 2016 Feb 22. PMID 26912555